CLINICAL TRIAL: NCT06004687
Title: Effects of Acetaminophen Preemptive Analgesia on Anesthesia Recovery Time and Postoperative Cognitive Function in Patients Undergoing Gastrointestinal Tumor Surgery
Brief Title: Effect of Acetaminophen Preemptive Analgesia on Postoperative Cognitive Function
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zhhszjjh
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Function
Keywords: acetaminophen mannitol; cognitive function; anesthesia recovery time; gastrointestinal tumor surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- By applying acetaminophen mannitol to patients with gastrointestinal tumors before surgery (Active Comparator): Acetaminophen mannitol injection 50ml(500mg) intravenously pumped 30 minutes before surgery
  Interventions: Drug: acetaminophen mannitol
- By applying normal saline to patients with gastrointestinal tumors before surgery (Placebo Comparator): Normal saline injection 50ml intravenously pumped 30 minutes before surgery
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: acetaminophen mannitol — Intravenous acetaminophen was administered 30 minutes before anesthesia
  Arms: By applying acetaminophen mannitol to patients with gastrointestinal tumors before surgery
Drug: Normal saline — Intravenous acetaminophen was administered 30 minutes before anesthesia
  Arms: By applying normal saline to patients with gastrointestinal tumors before surgery

SUMMARY:
Patients undergoing gastrointestinal tumor surgery are prone to delayed recovery and postoperative cognitive dysfunction due to greater trauma and longer operation time. Pre-analgesia can reverse the effects of nociceptive stimulation on recovery from general anesthesia and postoperative cognitive function. Intravenous injection of non-steroidal drugs can effectively reduce postoperative pain and the use of opioids. Therefore, This study selected acetaminophen mannitol injection for preemptive analgesia to observe the effects on anesthesia recovery time and postoperative cognitive function of patients undergoing gastrointestinal tumor surgery, providing new ideas for reducing cognitive dysfunction in patients undergoing gastrointestinal tumor surgery

DETAILED DESCRIPTION:
By administering acetaminophen to patients with gastrointestinal tumors before surgery, recording the time to recovery from anesthesia, and assessing cognitive function status by CAM on the first, third, and seventh day after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastrointestinal tumor surgery
* American Society of Anesthesiologists（ASA）≤Ⅲ

Exclusion Criteria:

* History of severe adverse reactions to oral acetaminophen
* Dysfunction of heart, liver, kidney and other important organs
* History of chronic pain
* Oral non-steroidal or opioid drugs
* Patients who do not accept clinical trials

Ages: 16 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | 1/3/7 days after the surgery
  The confusion assessment method (CAM) was used to assess postoperative cognitive dysfunction

SECONDARY OUTCOMES:
Recovery time | immediately after the surgery
  The postoperative recovery time was recorded

OTHER OUTCOMES:
Neurotransmitters in the blood | 1/3/7 days after the surgery
  Neurotransmitters include epinephrine, norepinephrine, and so on

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Chen, Study Chair — Chair
Locations (1):
- Affiliated Hospital of nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No